CLINICAL TRIAL: NCT03378531
Title: An Open-label, Multicentre Extension Study to Evaluate the Long-Term Safety, Tolerability and Effects of Intravenous AEB1102 in Patients With Arginase I Deficiency Who Previously Received Treatment in Study CAEB1102-101A
Brief Title: A Study of AEB1102 (Pegzilarginase) in Patients With Arginase I Deficiency
Acronym: AEB1102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-102A
Record Dates: First submitted 2017-12-11; First posted 2017-12-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arginase I Deficiency; Hyperargininemia
MeSH Terms: conditions — Hyperargininemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AEB1102 (Experimental): Each patient may receive AEB1102 administered IV for up to approximately 4 years.
  Interventions: Drug: AEB1102

INTERVENTIONS:
Drug: AEB1102 — modified human arginase I
  Other Names: Co-ArgI-PEG; Pegzilarginase

SUMMARY:
The purpose of this study is to investigate the long-term safety, tolerability, immunogenicity, pharmacokinetics and pharmacodynamics of intravenous AEB1102 in patients who complete Study CAEB1102-101A.

DETAILED DESCRIPTION:
Purpose of this study is to investigate the long-term safety, tolerability, immunogenicity, pharmacokinetics and pharmacodynamics of intravenous AEB1102 in patients who complete Study CAEB1102-101A.

ELIGIBILITY:
Inclusion Criteria:

1. Complete treatment in Study CAEB1102-101A without experiencing any clinically significant adverse event or other unmanageable drug toxicity that would preclude continued dosing
2. Confirmation by the Investigator and the Sponsor determine that it is acceptable for the patient to continue dosing with AEB1102
3. If female and of child-bearing potential, has a negative serum pregnancy test within 7 days before enrollment
4. If sexually active (male or female), must be surgically sterile, post-menopausal (female), or must agree to use a physician-approved method of birth control during the study and for a minimum of 30 days after the last study drug administration
5. Patient or legal guardian is able and willing to provide written informed consent and where required assent, and to comply with all requirements of study participation (including all study procedures and continuation of prescribed diet without modification), prior to any screening procedures

Exclusion Criteria:

1. Clinically significant concurrent disease, serious intercurrent illness, or other extenuating circumstances

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | up to 4 years
  Incidence of treatment-related adverse events

SECONDARY OUTCOMES:
Cmax Cmin | up to 4 years
  Cmax Cmin

CONTACTS AND LOCATIONS:
Overall Officials: Cortney Caudill, Study Director — Aeglea Biotherapeutics, Inc.
Locations (7):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - University of Florida, Gainesville, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UTSW, Dallas, Texas
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Centro Hospitalar S. Joao, Porto, Portugal
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Diaz GA, Schulze A, McNutt MC, Leao-Teles E, Merritt JL 2nd, Enns GM, Batzios S, Bannick A, Zori RT, Sloan LS, Potts SL, Bubb G, Quinn AG. Clinical effect and safety profile of pegzilarginase in patients with arginase 1 deficiency. J Inherit Metab Dis. 2021 Jul;44(4):847-856. doi: 10.1002/jimd.12343. Epub 2021 Jan 26. PMID 33325055